CLINICAL TRIAL: NCT03191942
Title: Variation of Orthokeratology Lens Treatment Zone (VOLTZ) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Pauline Cho, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20170118004
Record Dates: First submitted 2017-06-14; First posted 2017-06-19 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Myopia
Keywords: Myopia control; Orthokeratology; Children; Treatment zone
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified ortho-k lenses (Experimental): Participants wearing ortho-k lens with a modified BOZD of 5mm
  Interventions: Device: Modified ortho-k lenses
- Ortho-k lenses (Active Comparator): Participants wearing ortho-k lens with a standardized BOZD of 6mm
  Interventions: Device: Ortho-k lenses

INTERVENTIONS:
Device: Modified ortho-k lenses — KETT MC lens
  Arms: Modified ortho-k lenses
Device: Ortho-k lenses — KATT BeFree lens
  Arms: Ortho-k lenses

SUMMARY:
This project aims to study the effects of treatment characteristics on myopia control in orthokeratology by investigating the effects of modified treatment zone by reducing the lens back optic zone diameter on the effect of myopia control. The project will be a two-year randomized, double-masked (examiner - mask axial length only) study conducted at The Hong Kong Polytechnic University recruiting sixty Chinese subjects aged between 6-11. Subjects will be randomly assigned to two ortho-k groups. The Control group will wear KATT BeFree lens with a BOZD of 6mm while the Test group will wear KATT MC lens with a modified BOZD of 5mm.

DETAILED DESCRIPTION:
Orthokeratology (Ortho-k) treatment reduces the degree of myopia of the eye by flattening the central cornea. This central flattened zone is referred to as the treatment zone (TZ). Munnerlyn's formula describes the negative correlation between refractive correction and treatment zone size given a maximum ablation depth limited by the patient's corneal thickness in refractive surgery. This implies smaller TZ for higher myopic reduction and, indeed, a study found marginally smaller TZ of 0.3mm in higher myopic group. In ortho-k, it has been speculated that TZ may be associated with the effect of the treatment. The TZ is defined as the central flattened area enclosed by points with zero power/curvature changes comparing to pre-treatment condition on various topography maps.

Previous studies determine the TZ characteristics based on different types of topographical subtractive maps including tangential, axial and refractive maps. A study compared TZ parameters derived from the three different maps. The study defined the TZ as the area enclosed by zero power change in different subtractive maps; 12 such points equally spaced 30 degree apart to construct a best-fit ellipse. Geometrical center of this ellipse was used to determine the TZ decentration and TZ diameter along vertical and horizontal axes. The study found significantly less TZ decentration and diameter in tangential map comparing to axial and refractive maps and no significant difference between the latter two. Based on these findings, the investigators suggested that either refractive or axial map would be of high validity and accuracy in determining TZ characteristics.

The current study would investigate the effect of TZ on myopic control in ortho-k. TZ, defined as the area enclosed by zero power change in subjective maps will be employed. The tangential and refractive subtractive maps will be used to determine the TZ. Characteristics of the TZ, including diameter, slope, depth, volume, would be analyzed based on topographical subtractive maps and the effect of each of these characteristics on myopia control will be evaluated. The role of pupil size during normal viewing condition (distance and near) will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Manifest myopia between 1.00-4.00D in both eyes at screening visit
* Manifest astigmatism ≤2.50D; with-the-rule astigmatism (axes 180 ± 30)

  * 2.50D; astigmatism with other axes ≤0.50D in both eyes at screening visit
* <1.00D difference in manifest spherical equivalent (SE) between the two eyes at screening visit
* Baseline cycloplegic objective refraction between 1.00-4.00D in sphere; astigmatism ≤2.50D; <1.00D difference in manifest SE between the two eyes
* Best-corrected logMAR visual acuity 0.10 or better in both eyes Symmetrical corneal topography with corneal toricity <2.00D in either eye
* Normal ocular health other than myopia
* Agree to be randomized and to attend the scheduled visits and aftercare

Exclusion Criteria:

* Contraindications to atropine: known allergies or cardiovascular disease, epilepsy
* Contraindications to contact lens wear and ortho-k: corneal scar, history of ocular inflammation/infection, limbus-to-limbus corneal cylinder and dislocated corneal apex
* Strabismus or amblyopia
* History of myopia control treatment (e.g. soft contact lenses, progressive add spectacles, atropine eye drops)
* Rigid contact lens (including ortho-k) wear experience
* Systemic condition which might affect refractive development (for example, Down syndrome, Marfan's syndrome)
* Ocular conditions which might affect refractive error (for example, cataract, ptosis)
* Poor response to lens wear including poor lens handling, poor vision and/ocular response after lens modifications
* Poor compliance with schedule visits

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2021-03-21 (Actual); Study Completion 2021-07-27 (Actual)

PRIMARY OUTCOMES:
Change in axial length before and after two years of lens wear | 2 years
  To determine the change in axial length measured at baseline and two years after lens wear using IOLMaster

SECONDARY OUTCOMES:
Treatment zone characteristics | 2 years
  Corneal topography will be determined by Medmont topographer and the treatment zone characteristics will be determined from the subtractive maps
Pupil sizes | 2 years
  Photopic and mesotopic pupil sizes
Choroidal thickness | 2 years
  Choroidal thickness measurement will be determined by both LenStar and posterior OCT

CONTACTS AND LOCATIONS:
Overall Officials: Pauline Cho, phd, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - School of Optometry, The Hong Kong Polytechnic University, Kowloon
  - School of Optometry, Kowloon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Owens H, Garner LF, Craig JP, Gamble G. Posterior corneal changes with orthokeratology. Optom Vis Sci. 2004 Jun;81(6):421-6. doi: 10.1097/01.opx.0000135097.99877.5d. PMID 15201715
- [Background] Lu F, Simpson T, Sorbara L, Fonn D. The relationship between the treatment zone diameter and visual, optical and subjective performance in Corneal Refractive Therapy lens wearers. Ophthalmic Physiol Opt. 2007 Nov;27(6):568-78. doi: 10.1111/j.1475-1313.2007.00520.x. PMID 17956362
- [Background] Gifford P, Swarbrick HA. The effect of treatment zone diameter in hyperopic orthokeratology. Ophthalmic Physiol Opt. 2009 Nov;29(6):584-92. doi: 10.1111/j.1475-1313.2009.00672.x. Epub 2009 Aug 3. PMID 19663928
- [Background] Tahhan N, Du Toit R, Papas E, Chung H, La Hood D, Holden AB. Comparison of reverse-geometry lens designs for overnight orthokeratology. Optom Vis Sci. 2003 Dec;80(12):796-804. doi: 10.1097/00006324-200312000-00009. PMID 14688542
- [Background] Sridharan R, Swarbrick H. Corneal response to short-term orthokeratology lens wear. Optom Vis Sci. 2003 Mar;80(3):200-6. doi: 10.1097/00006324-200303000-00009. PMID 12637831
- [Background] Munnerlyn CR, Koons SJ, Marshall J. Photorefractive keratectomy: a technique for laser refractive surgery. J Cataract Refract Surg. 1988 Jan;14(1):46-52. doi: 10.1016/s0886-3350(88)80063-4. PMID 3339547
- [Derived] Guo B, Cho P, Cheung SW, Kojima R, Vincent S. Optical changes and association with axial elongation in children wearing orthokeratology lenses of different back optic zone diameter. Eye Vis (Lond). 2023 Jul 1;10(1):25. doi: 10.1186/s40662-023-00344-3. PMID 37391828